CLINICAL TRIAL: NCT01136746
Title: Randomized Clinical Trial of Subcutaneous Analog Basal Bolus Therapy Versus Sliding Scale Human Regular Insulin in the Hospital Management of Hyperglycemia in Non-Critically Ill Patients Without Known History of Diabetes: The HMH Trial
Brief Title: Hospital Management of Hyperglycemia Study of Insulin Glargine Plus Insulin Lispro Versus Human Regular Insulin
Acronym: HMH
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13698; F3Z-US-IOPZ (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-06-02; First posted 2010-06-03 (Estimated); Results first posted 2012-10-12 (Estimated); Last update posted 2012-11-13 (Estimated); Status verified 2012-11

CONDITIONS: Hyperglycemia
Keywords: Hyperglycemia; Diabetes; Hospital; Diabetic
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus | interventions — Insulin; Insulin Lispro; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sliding scale regular insulin (Active Comparator)
  Interventions: Drug: Human regular insulin
- Basal-bolus therapy (Experimental)
  Interventions: Drug: Insulin lispro; Drug: Insulin glargine

INTERVENTIONS:
Drug: Human regular insulin — Administered subcutaneously, four times daily, according to sliding scale insulin algorithm throughout hospital study period (1 to 10 days post-randomization)
  Other Names: Humulin R; LY041001
  Arms: Sliding scale regular insulin
Drug: Insulin lispro — Administered subcutaneously, 3 to 4 times daily, according to plasma glucose levels throughout hospital study period (1 to 10 days post-randomization)
  Other Names: Humalog; LY275585
  Arms: Basal-bolus therapy
Drug: Insulin glargine — Administered subcutaneously, once daily, according to plasma glucose levels throughout hospital study period (1 to 10 days post-randomization)
  Other Names: Lantus
  Arms: Basal-bolus therapy

SUMMARY:
The purpose of this study is to compare the use of insulin glargine plus insulin lispro to human regular insulin for treatment of hyperglycemia in the hospital setting in patients without known prior history of diabetes.

DETAILED DESCRIPTION:
This study involves a comparison of 2 methods for administering subcutaneous insulin therapy to non-critically ill adult patients with hyperglycemia and without known history of diabetes who are admitted to non-intensive care unit (ICU) general medical hospital services. Basal-bolus therapy, considered the gold standard for glucose control in patients with known diabetes, will be compared with sliding scale insulin, a commonly used method of glucose control (prevailing standard practice) in hospitalized patients. In this study, basal-bolus therapy will consist of once-daily glargine plus lispro 3 to 4 times daily adjusted to achieve pre-meal capillary plasma glucose <140 milligrams per deciliter (mg/dL) and bedtime capillary plasma glucose <180 mg/dL for patients who are eating [predose plasma glucose <140 mg/dL for patients with nil per os (NPO) orders]; sliding scale insulin will be administered using human regular insulin 4 times daily as needed adjusted to achieve predose capillary plasma glucose target <140 mg/dL in patients who are eating or have NPO orders.

ELIGIBILITY:
Major Inclusion Criteria:

* No known history of diabetes
* Admission or pre-entry plasma glucose (PG) level between 140 and 400 mg/dL
* Non-critically ill and admitted to acute care medical services
* Have a body mass index greater than or equal to 18.5 kg/m^2 and less than or equal to 45 kilograms per square meter (kg/m^2)

Major Exclusion Criteria:

* Received any insulin/analog therapy for longer than 108 hours prior to study entry or intermediate- or long-acting insulin/analogs (neutral protamine Hagedorn, detemir, or glargine) in the 24 hours prior to randomization or any intravenous insulin therapy prior to randomization
* Laboratory evidence of diabetic ketoacidosis for patients with pre-randomization PG greater than 250 mg/dL
* Have taken any oral or injectable antihyperglycemic medications other than insulin within 3 months prior to study entry
* Have acute critical illness or are expected to require admission to an ICU or equivalent or be treated with glucocorticoid therapy during the hospital study period
* Expected hospitalization less than 24 hours post-randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-03; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (12):
- United States (12):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Weston, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Topeka, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hazard, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangor, Maine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kansas City, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee

REFERENCES:
- [Background] Workgroup on Hypoglycemia, American Diabetes Association. Defining and reporting hypoglycemia in diabetes: a report from the American Diabetes Association Workgroup on Hypoglycemia. Diabetes Care. 2005 May;28(5):1245-9. doi: 10.2337/diacare.28.5.1245. No abstract available. PMID 15855602
- [Background] American Diabetes Association. Standards of medical care in diabetes--2010. Diabetes Care. 2010 Jan;33 Suppl 1(Suppl 1):S11-61. doi: 10.2337/dc10-S011. No abstract available. PMID 20042772
- [Background] Moghissi ES, Korytkowski MT, DiNardo M, Einhorn D, Hellman R, Hirsch IB, Inzucchi SE, Ismail-Beigi F, Kirkman MS, Umpierrez GE; American Association of Clinical Endocrinologists; American Diabetes Association. American Association of Clinical Endocrinologists and American Diabetes Association consensus statement on inpatient glycemic control. Endocr Pract. 2009 May-Jun;15(4):353-69. doi: 10.4158/EP09102.RA. No abstract available. PMID 19454396
- [Background] Umpierrez GE, Smiley D, Zisman A, Prieto LM, Palacio A, Ceron M, Puig A, Mejia R. Randomized study of basal-bolus insulin therapy in the inpatient management of patients with type 2 diabetes (RABBIT 2 trial). Diabetes Care. 2007 Sep;30(9):2181-6. doi: 10.2337/dc07-0295. Epub 2007 May 18. PMID 17513708
- [Background] Umpierrez GE, Hor T, Smiley D, Temponi A, Umpierrez D, Ceron M, Munoz C, Newton C, Peng L, Baldwin D. Comparison of inpatient insulin regimens with detemir plus aspart versus neutral protamine hagedorn plus regular in medical patients with type 2 diabetes. J Clin Endocrinol Metab. 2009 Feb;94(2):564-9. doi: 10.1210/jc.2008-1441. Epub 2008 Nov 18. PMID 19017758

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Started | 9 | 7
Completed | 6 | 4
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol Violation | 2 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy | Total
Number analyzed (Participants) | 9 | 7 | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 60.2 (16.8) | 51.4 (8.5) | 56.4 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 8 | 7 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Mean Plasma Glucose (MPG) Throughout Hospital Study Period
Description: Overall MPG is derived as the mean of plasma glucose (PG) readings from Day/Visit 1 to Day/Visit 10.
Time Frame: Throughout hospital study period (1 to 10 days post-randomization)
Population: All randomized participants who had at least one post-baseline glucose measurement.
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Number analyzed (Participants) | 9 | 6
milligrams per deciliter (mg/dL) | 167.6 (48.5) | 128.4 (22.4)

2. Primary Outcome: Percentage of Capillary Plasma Glucose Measurements Within the Range of 71 to 179 mg/dL Throughout the Hospital Study Period
Description: Results are reported as the percentage of total number of capillary plasma glucose measurements within the range of 71 to 179 mg/dL for each treatment arm.
Time Frame: Throughout hospital study period (1 to 10 days post-randomization)
Population: All randomized participants who had at least one post-baseline glucose measurement.
Measure: Number; unit: percentage of capillary PG measurements
Units Other Than Participants: capillary plasma glucose measurements
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Number analyzed (Participants) | 9 | 6
Number analyzed (capillary plasma glucose measurements) | 70 | 51
percentage of capillary PG measurements | 81.4 | 84.3

3. Secondary Outcome: Mean Plasma Glucose (MPG) by Hospital Day
Description: The intent was to report results up to Day 10; however, due to low enrollment, mean and standard deviations are only reported up to Day 7.
Time Frame: Day 1 up to day 7 of hospital study period
Population: All randomized participants who had at least one post-baseline glucose measurement and a plasma glucose measurement at specified timepoint.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Number analyzed (Participants) | 9 | 6
mg/dL
  Day 1 (n=6, n=6) | 178.1 (54.9) | 149.9 (17.2)
  Day 2 (n=8, n=5) | 175.2 (57.9) | 124.0 (29.8)
  Day 3 (n=6, n=3) | 151.0 (46.9) | 128.5 (28.5)
  Day 4 (n=2, n=1) | 132.5 (2.12) | 96.3 (NA) — Standard Deviation cannot be calculated when there is only one participant.
  Day 5 (n=1, n=1) | 154.8 (NA) — Standard Deviation cannot be calculated when there is only one participant. | 104.6 (NA) — Standard Deviation cannot be calculated when there is only one participant.
  Day 6 (n=1, n=1) | 138.0 (NA) — Standard Deviation cannot be calculated when there is only one participant. | 111.0 (NA) — Standard Deviation cannot be calculated when there is only one participant.
  Day 7 (n=0, n=1) | NA (NA) — Cannot calculate a Mean or Standard Deviation with zero participants. | 108.0 (NA) — Standard Deviation cannot be calculated when there is only one participant.

4. Secondary Outcome: Percentage of Plasma Glucose Measurements Within Range 71 to 179 mg/dL by Hospital Day
Description: Due to low enrollment, this outcome measure was not analyzed.
Time Frame: Day 1 up to day 10 of hospital study period
Population: Due to low enrollment, zero participants were analyzed.
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage of Participants Achieving MPG Within Range 71 to 179 mg/dL and Within the Target of 100 to 179 mg/dL Throughout Hospital Study Period
Description: Due to low enrollment, this outcome measure was not analyzed.
Time Frame: Throughout hospital study period (1 to 10 days post-randomization)
Population: Due to low enrollment, zero participants were analyzed.
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percentage of Participants Achieving MPG Within Range 71 to 179 mg/dL and Within the Target of 100 to 179 mg/dL by Hospital Day
Description: Due to low enrollment, this outcome measure was not analyzed.
Time Frame: Day 1 up to day 10 of hospital study period
Population: Due to low enrollment, zero participants were analyzed.
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Mean Fasting Plasma Glucose (FPG) by Hospital Day
Description: Due to low enrollment, this outcome measure was not analyzed.
Time Frame: Day 1 up to day 10 of hospital study period
Population: Due to low enrollment, zero participants were analyzed.
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Mean FPG Throughout Hospital Study Period
Description: Due to low enrollment, this outcome measure was not analyzed.
Time Frame: Throughout hospital study period (1 to 10 days post-randomization)
Population: Due to low enrollment, zero participants were analyzed.
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Percentage of Fasting Capillary PG Measurements Within the Range of 71 to 139 mg/dL and Within the Target of 100 to 139 mg/dL Throughout the Hospital Study Period
Description: Due to low enrollment, this outcome measure was not analyzed.
Time Frame: Throughout the hospital study period (1 to 10 days post-randomization)
Population: Due to low enrollment, zero participants were analyzed.
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Percentage of Fasting Capillary PG Measurements Within the Range of 71 to 139 mg/dL and Within the Target of 100 to 139 mg/dL by Hospital Day
Description: Due to low enrollment, this outcome measure was not analyzed.
Time Frame: Day 1 up to day 10 of hospital study period
Population: Due to low enrollment, zero participants were analyzed.
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Percentage of Participants Achieving Mean FPG Range of 71 to 139 mg/dL and Target of 100 to 139 mg/dL Throughout the Hospital Study Period
Description: Due to low enrollment, this outcome measure was not analyzed.
Time Frame: Throughout the hospital study period (1 to 10 days post-randomization)
Population: Due to low enrollment, zero participants were analyzed.
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Percentage of Participants Achieving Mean FPG Range of 71 to 139 mg/dL and Target of 100 to 139 mg/dL by Hospital Day
Description: Due to low enrollment, this outcome measure was not analyzed.
Time Frame: Day 1 up to day 10 of hospital study period
Population: Due to low enrollment, zero participants were analyzed.
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Percentage of Capillary PG Measurements >240 mg/dL Throughout the Hospital Study Period
Description: Due to low enrollment, this outcome measure was not analyzed.
Time Frame: Throughout the hospital study period (1 to 10 days post-randomization)
Population: Due to low enrollment, zero participants were analyzed.
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Number analyzed (Participants) | 0 | 0

14. Secondary Outcome: Percentage of Capillary PG Measurements >240 mg/dL by Hospital Day
Description: Due to low enrollment, this outcome measure was not analyzed.
Time Frame: Day 1 up to day 10 of hospital study period
Population: Due to low enrollment, zero participants were analyzed.
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Total Daily Dose (TDD) of Insulin (Units) Throughout the Hospital Study Period
Description: Due to low enrollment, this outcome measure was not analyzed.
Time Frame: Throughout the hospital study period (1 to 10 days post-randomization)
Population: Due to low enrollment, zero participants were analyzed.
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: TDD of Insulin (Units/kg) Throughout the Hospital Study Period
Description: Due to low enrollment, this outcome measure was not analyzed.
Time Frame: Throughout the hospital study period (1 to 10 days post-randomization)
Population: Due to low enrollment, zero participants were analyzed.
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: TDD of Insulin (Units) by Hospital Day
Description: Due to low enrollment, this outcome measure was not analyzed.
Time Frame: Day 1 up to day 10 of hospital study period
Population: Due to low enrollment, zero participants were analyzed.
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: TDD of Insulin (Units/kg) by Hospital Day
Description: Due to low enrollment, this outcome measure was not analyzed.
Time Frame: Day 1 up to day 10 of hospital study period
Population: Due to low enrollment, zero participants were analyzed.
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Length of Hospital Stay Post-randomization Throughout the Hospital Study Period
Description: Due to low enrollment, this outcome measure was not analyzed.
Time Frame: Throughout the hospital study period (1 to 10 days post-randomization)
Population: Due to low enrollment, zero participants were analyzed.
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Number (Incidence) of Hypoglycemia and Severe Hypoglycemia Episodes, Throughout Hospital Study Period
Description: Hypoglycemia was defined as any time a recorded capillary PG level is ≤70 mg/dL, even if it is not associated with signs or symptoms, or treatment consistent with current guidelines (ADA 2005; ADA 2010). Severe hypoglycemia was defined as an episode associated with a recorded capillary (or venous) PG <40 mg/dL (Umpierrez et al. 2007; Moghissi et al. 2009; Umpierrez et al. 2009), even if it is not associated with need for assistance or neuroglycopenic symptoms (ADA 2005) or prompt recovery after oral carbohydrate, glucagon, or IV glucose.
Time Frame: Throughout hospital study period (1 to 10 days post-randomization)
Population: All randomized participants who had at least one post-baseline glucose measurement.
Measure: Number; unit: hypoglycemic episodes
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Number analyzed (Participants) | 9 | 6
hypoglycemic episodes
  Hypoglycemic Episodes | 1 | 3
  Severe Hypoglycemic Episodes | 0 | 0

21. Secondary Outcome: Number of Hypoglycemia and Severe Hypoglycemia Episodes Adjusted for 30 Days (Rate), Throughout Hospital Study Period
Description: Hypoglycemia was defined as any time a recorded capillary PG level is ≤70 mg/dL, even if it is not associated with signs or symptoms, or treatment consistent with current guidelines (ADA 2005; ADA 2010). Severe hypoglycemia was defined as an episode associated with a recorded capillary (or venous) PG <40 mg/dL, even if it is not associated with need for assistance or neuroglycopenic symptoms (ADA 2005) or prompt recovery after oral carbohydrate, glucagon, or IV glucose. Due to low enrollment, this outcome measure was not analyzed.
Time Frame: Throughout hospital study period (1 to 10 days post-randomization)
Population: Due to low enrollment, zero participants were analyzed.
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Number (Incidence) of Hypoglycemia and Severe Hypoglycemia Episodes, by Hospital Day
Description: as for outcome 21
Time Frame: Day 1 up to day 10 of hospital study period
Population: Due to low enrollment, zero participants were analyzed.
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Number of Hypoglycemia and Severe Hypoglycemia Episodes Adjusted for 30 Days (Rate), by Hospital Day
Description: as for outcome 21
Time Frame: Day 1 up to day 10 of hospital study period
Population: Due to low enrollment, zero participants were analyzed.
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events Throughout Hospital Study Period
Description: Treatment-emergent adverse event - any untoward medical occurrence that either occurred or worsened at any time after treatment baseline and which did not necessarily have a causal relationship with this treatment. A summary of adverse events is located in the Reported Adverse Event Module.
Time Frame: Throughout hospital study period (1 to 10 days post-randomization)
Population: All randomized participants
Measure: Number; unit: participants
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Number analyzed (Participants) | 9 | 7
participants | 1 | 2

25. Secondary Outcome: Percentage of Participants Requiring Intensive Care Unit Transfer
Description: Due to low enrollment, this outcome measure was not analyzed.
Time Frame: Throughout hospital study period (1 to 10 days post-randomization)
Population: Due to low enrollment, zero participants were analyzed.
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Number analyzed (Participants) | 0 | 0

26. Secondary Outcome: Percentage of Participants With Deterioration of Renal Function Throughout the Hospital Study Period
Description: Deterioration of renal function was defined by an increase in serum creatinine by >0.5 milligrams per deciliter (mg/dL). Due to low enrollment, this outcome measure was not analyzed.
Time Frame: Throughout hospital study period (1 to 10 days post-randomization)
Population: Due to low enrollment, zero participants were analyzed.
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Percentage of Participants With Documented Nosocomial Infections
Description: Due to low enrollment, this outcome measure was not analyzed.
Time Frame: Throughout hospital study period (1 to 10 days post-randomization)
Population: Due to low enrollment, zero participants were analyzed.
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Number of Participants With Major Adverse Cardiovascular Events (MACE)
Description: MACE was defined as the composite of all-cause death, nonfatal myocardial infarction (MI), or nonfatal stroke. Due to low enrollment, this outcome measure was not analyzed.
Time Frame: Throughout hospital study period (1 to 10 days post-randomization)
Population: Due to low enrollment, zero participants were analyzed.
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Sliding Scale Regular Insulin | Basal-bolus Therapy
Serious Adverse Events (participants affected / at risk) | 1/9 | 0/7
Other Adverse Events (participants affected / at risk) | 1/9 | 2/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sliding Scale Regular Insulin (N=9) | Basal-bolus Therapy (N=7)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sliding Scale Regular Insulin (N=9) | Basal-bolus Therapy (N=7)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
High density lipoprotein decreased (Investigations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to low enrollment, this trial was terminated early, leading to small numbers of participants analyzed or some outcome measures not being able to be analyzed at all.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days